CLINICAL TRIAL: NCT02692638
Title: Prospective, Randomized Trial Comparing Early Laparoscopic Enterolysis Versus a Time-limited Trial of Nonoperative Management for High-grade Small Bowel Obstruction
Brief Title: Trial Comparing Early Laparoscopic Enterolysis Versus Nonoperative Management for High-grade SBO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low enrollment; PI left institution
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1512016944
Record Dates: First submitted 2016-02-15; First posted 2016-02-26 (Estimated); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Small Bowel Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early laparoscopic enterolysis (Experimental): Patient randomized to the early laparoscopy arm will undergo diagnostic laparoscopy within 24 hours of admission (depending on surgeon and operating room availability). Standard laparoscopy will be performed including supine positioning, sequential compression devices, and appropriate pre-incision antibiotics. Trocar placement will be at the surgeon's discretion and as appropriate for the patient's previous incisions. The necessity for conversion will be left to the discretion of the attending surgeon. Post operative management will conform to the standards of care. Nasogastric tubes will not be routinely placed.
  Interventions: Procedure: Early laparoscopic enterolysis
- trial of nonoperative management (Active Comparator): Patients randomized to the trial of nonoperative management arm will undergo standard therapy including nil per os (NPO), nasogastric decompression only if actively vomiting, intravenous fluids while awaiting return of bowel function. Patients who do not achieve return of bowel function within 72 hours of admission will undergo attempted laparoscopic enterolysis with the understanding that conversion to open procedure may be necessary.
  Interventions: Procedure: nonoperative management

INTERVENTIONS:
Procedure: Early laparoscopic enterolysis — The surgeon will make about 3-4 small incisions in the participant's abdomen. A port (nozzle) is inserted into one of the slits, and carbon dioxide gas inflates the abdomen. A laparoscope is inserted through another port. The laparoscope looks like a telescope with a light and camera on the end so the surgeon can see inside the abdomen. Surgical instruments are placed in the other small openings and used to cut the scar tissue in order to relieve the obstruction. After all this has been accomplished, the carbon dioxide is released out of the abdomen through the slits, and then these sites are closed with sutures or staples, or covered with glue-like bandage and steri-strips.
  Arms: Early laparoscopic enterolysis
Procedure: nonoperative management — Sometimes a bowel obstruction can be treated by suctioning out the contents of the stomach, giving IV fluids, and not letting the patient eat for a few days.
  Arms: trial of nonoperative management

SUMMARY:
The goal is to assess the appropriateness of the standard practice of a trial of nonoperative management for high grade small bowel obstruction (currently up to 72 hours based on available literature). The investigator will offer early laparoscopic enterolysis (within 24 hours of admission) as the comparator group.

DETAILED DESCRIPTION:
Small bowel obstruction is a common disorder without a clearly superior management strategy. There are an estimated 300,000 surgeries performed annually with a health care expenditure burden in excess of 2.8 billion dollars. The investigators propose a new management paradigm including early laparoscopic management.

Contemporary management of SBO includes a trial of nonoperative management (TNOM) reportedly with resolution in upwards of 70% of patients.

Although it is one of the most common diagnosis for surgical admissions, there are few prospective, clinical trials to address the question surgical timing. Additionally, there are no prospective, randomized trials comparing early laparoscopy versus TNOM for high grade SBO. The hypothesis is that early laparoscopic enterolysis will result in decreased overall complications, shorter length of stay, decreased health care cost, and lower conversion rate to open laparotomy.

ELIGIBILITY:
Inclusion Criteria:

* CT A/P showing high grade obstruction (all patients will obtain a CT A/P as per Level 1 recommendations based on EAST practice guidelines) .
* High grade bowel obstruction is defined as:

  * Transition point
  * Distal small collapse with proximal dilatation
  * Small bowel feces sign
  * 50% difference in caliber change between proximal dilated bowel and distal decompressed bowel
  * Intra-abdominal free fluid without clinical signs of ischemia

Exclusion Criteria:

* Hemodynamic instability (SBP<90)
* Peritonitis
* Enterocutaneous fistula
* Cirrhosis
* previous enterolysis (more than 1)
* Contraindication to laparoscopic surgery
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-02-02 (Actual); Primary Completion 2016-10-13 (Actual); Study Completion 2016-10-13 (Actual)

PRIMARY OUTCOMES:
Number of complications (per National Surgical Quality Improvement Project) | 2 weeks
  complications counted : Superficial surgical site infection (SSI), Deep SSI, Organ space SSI, Wound disruption, pneumonia, Pulmonary embolism, ventilator days, Acute Kidney Injury (AKI), Acute renal failure (ARF), Urinary Tract Infection (UTI), Stroke, Cardiac arrest, Myocardial Infarction (MI), Sepsis, Deep vein thrombosis (DVT)

SECONDARY OUTCOMES:
Average Length of stay | length of hospital stay, Time 0 is at randomization with expected length of stay less than 3 weeks.
  length, in days, of hospital stay, calculated by subtracting date of randomization from date of discharge
Average cost in dollars | length of hospital stay, Time 0 is at randomization with expected length of stay less than 3 weeks.
  average cost of care of patients per arm for length of hospital stay
number of subjects with hospital readmission | within 2 weeks of discharge
number of subjects with unplanned return to operating room | within two weeks of discharge
number of subjects with 30 day mortality | 30 days post operation

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Pei, MD, Principal Investigator — Yale University; Kimberly Davis, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No